CLINICAL TRIAL: NCT01102140
Title: The Impact of Pomegranate (Punica Granatum) Polyphenol Extract on Oxidative Stress, Ventricular Remodeling and Endothelial Function in Chronic Cardiomyopathy Complicated by Renal Insufficiency (ImPrOVE): a Pilot Study
Brief Title: The Impact of Pomegranate Extract on Chronic Cardiomyopathy Complicated by Renal Insufficiency (ImPrOVE): a Pilot Study
Acronym: ImPrOVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left University of Michigan
Sponsor: Jennifer Cowger , MD, MS (Other)
Collaborators: POM Wonderful LLC (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Cowger , MD, MS, Assistant Professor, study PI, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMPROVEHF
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Cardiomyopathy; Heart Failure
Keywords: Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Cardiomyopathies; Heart Failure | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will either receive POMx or matching placebo (sugar pill)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- POMx (Active Comparator): 15 subjects will received 1000 mg of oral POMx for 12 weeks.
  Interventions: Drug: POMx, pomegranate polyphenol extract
- Control- sugar Pill (Placebo Comparator): 15 subjects will receive a matching sugar pill for 12 weeks.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: POMx, pomegranate polyphenol extract — 1000 mg orally once daily.
  Arms: POMx
Drug: Sugar Pill — Matching sugar pill
  Arms: Control- sugar Pill

SUMMARY:
This blinded, controlled study will examine the impact of pomegranate polyphenol extract (POMx, from Pom Wonderful, LLC), 1000mg on cardiomyopathy in subjects with chronic renal insufficiency.

DETAILED DESCRIPTION:
Heart failure (HF) is a disease of great prevalence in the U.S. with an associated high morbidity and mortality. In individuals with concomitant chronic renal insufficiency (CRI), outcomes are even worse due to pharmaceutical under treatment and higher baseline levels of oxidative stress. Reactive oxygen species (ROS) are generated during mechanoenergetic uncoupling and can cause myocardial protein, lipid, and DNA damage, leading to the development of HF. One means of preventing the progression of HF may be through ROS reduction or an improvement in systemic or local oxidative stress handling. In this randomized, single blind placebo-controlled pilot study, we hypothesize that 12 weeks of treatment with oral pomegranate extract (POMx) will lead to a reduction in oxidative stress (as assessed by measuring thiobarbituric acid-reactive substances, F8-isoprostanes, and glutathione) in subjects (n=30) with cardiomyopathy (LVEF ≤40%) and CRI (GFR <60 ml/hr). Secondary aims include assessing the impact of POMx on myocardial remodeling and endothelial dysfunction by measuring serum collagen levels and asymmetric dimethylarginine, respectively. Findings from this study will serve as pilot data for a larger randomized trial of longer term POMx therapy in subjects with cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥21 years of age) with cardiomyopathy (ejection fraction ≤40%) of at least 1 year duration and CRI (GFR <60 cc/hr for at least 3 months) will be eligible for enrollment.
* Subjects must have New York Heart Association (NYHA) functional class I-III symptoms and be on stable doses of HF evidence-based therapies (β-blocker, ACE inhibitor or ARBs, aldosterone inhibitor [if appropriate]) for at least 3 months or have a documented contraindication or intolerance to such therapy

Exclusion Criteria:

* Subjects admitted to a hospital for acute myocardial infarction (defined as positive troponins) or HF exacerbation within the last 6 months will not be eligible for enrollment.
* Subjects on warfarin or rosuvastatin will also be excluded.
* Other exclusion criteria are as follows:

  * HF that is deemed to be congenital or infiltrative in etiology
  * the presence of a life-threatening illness with a projected survival ≤6 months; ongoing infection
  * pregnancy
  * inability to follow-up
  * end-stage renal disease requiring dialysis
  * renal transplant listing
  * recent (within last 6 months) POMx use or intake >8 ounces daily of pomegranate juice
  * known hypersensitivity to any fruit in the Punicaceae family
  * connective tissue or collagen vascular disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Matthews, MD, MS, Principal Investigator — Univeristy of Michigan Health System; Bertram Pitt, MD, Study Chair — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- POMx: The POMx subjects received 1000 mg of oral POMx for 12 weeks.
  POMx, pomegranate polyphenol extract: 1000 mg orally once daily.
- Control- Sugar Pill: The control subjects received a matching sugar pill for 12 weeks.
  Sugar Pill: Matching sugar pill
Period: Overall Study
Arm/Group | POMx | Control- Sugar Pill
Started | 13 | 7
Completed | 10 | 5
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Investigator terminated study | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | POMx | Control- Sugar Pill | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 3 | 2 | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [49 to 64] | 58 [52 to 64] | 57 [50 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 13 | 5 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 6 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Thiobarbituric Reactive Substances (TBARS)
Description: This is a serum marker of oxidative stress.
Time Frame: baseline and after 12 weeks
Population: Serum samples were obtained and frozen but never analyzed to obtain isoprostane values due to PI departure from study center prior to any batches being sent for analysis.
Arm/Group | POMx | Control- Sugar Pill
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: F-8 Isoprostanes
Description: This is a serum marker of oxidative stress.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Arm/Group | POMx | Control- Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Procollagen Types I (PINP) and III (PIIINP)
Description: This is a serum marker of collagen turnover (fibrosis/scar formation).
Time Frame: baseline and 12 weeks
Population: Serum samples were obtained and frozen but never analyzed to obtain procollagen values due to PI departure from study center prior to any batches being sent for analysis
Groups:
- POMx: The POMx subjects will receive 1000 mg of oral POMx for 12 weeks.
  POMx, pomegranate polyphenol extract: 1000 mg orally once daily.
Arm/Group | POMx | Control- Sugar Pill
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Asymmetric Dimethylarginine (ADMA)
Description: ADMA is a serum enzyme involved in metabolism of endothelium derived nitric oxide (NO). NO's has an important role in maintaining endothelial homeostasis. Elevated ADMA levels suggest impaired endothelial function.
Time Frame: baseline and 12 weeks
Population: Serum samples were obtained and frozen but never analyzed to obtain ADMA values due to PI departure from study center prior to any batches being sent for analysis
Arm/Group | POMx | Control- Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- POMx: 15 subjects received 1000 mg of oral POMx for 12 weeks.
  POMx, pomegranate polyphenol extract: 1000 mg orally once daily.
Arm/Group | POMx | Control- Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No